CLINICAL TRIAL: NCT01874444
Title: Verify the Effectiveness rTMS Using MEG
Acronym: rTMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TN2447
Record Dates: First submitted 2013-06-04; First posted 2013-06-11 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2013-12

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active rTMS1 (Experimental): Combined low frequency frontal and temporal repetitive transcranial magnetic stimulation of left primary auditory cortex and left dorsolateral prefrontal cortex .
  Interventions: Device: 1
- Active rTMS2 (Experimental): Temporal low frequency rTMS of left primary auditory cortex.
  Interventions: Device: 2
- Active rTMS3 (Experimental): Frontal low frequency rTMS of left dorsolateral prefrontal cortex .
  Interventions: Device: 3
- Sham rTMS4 (Sham Comparator): sham treatment Sham rTMS, applied with the same combination of parameters as active rTMS, except for the number of stimulations per session.
  Interventions: Device: 4

INTERVENTIONS:
Device: 1 — repetitive transcranial magnetic stimulation (Figured 8-Coil MCF-B65): 1000 stimuli of 1Hz rTMS over the left DLPFC (110% motor threshold) followed by 2000 stimuli of 1 Hz rTMS over the left temporal cortex (110% motor threshold), each consisting of 4 days of rTMS treatment. Participants will have an MRI scan and MEG recoding at the performed a week before rTMS. And MEG recording after 7day the application of rTMS
  Arms: Active rTMS1
Device: 2 — repetitive transcranial magnetic stimulation (Figured 8-Coil MCF-B65): 3000 stimuli of 1 Hz rTMS over the left temporal cortex (110% motor threshold), each consisting of 4 days of rTMS treatment.
  Participants will have an MRI scan and MEG recoding at the performed a week before rTMS. And MEG recording after 7day the application of rTMS.
  Arms: Active rTMS2
Device: 3 — repetitive transcranial magnetic stimulation (Figured 8-Coil MCF-B65): 3000 stimuli of 1 Hz rTMS over the left frontal cortex (110% motor threshold) each consisting of 4 days of rTMS treatment.
  Participants will have an MRI scan and MEG recoding at the performed a week before rTMS. And MEG recording after 7day the application of rTMS.
  Arms: Active rTMS3
Device: 4 — Sham rTMS, applied with the same combination of parameters as active rTMS, except for the number of stimulations per session.
  Participants will have an MRI scan and MEG recoding at the performed a week before rTMS. And MEG recording after 7day the application of rTMS.
  Arms: Sham rTMS4

SUMMARY:
The purpose of this study is to determine whether rTMS are effective in the treatment of tinnitus

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) of the dorsolateral prefrontal cortex (DLPFC) has an add-on effect for primary auditory cortex rTMS in improving tinnitus-related distress. We aimed to investigate whether rTMS of the dorsolateral prefrontal cortex and primary auditory cortex are capable of reducing tinnitus loudness. Linked to a neuronavigation system that is guided by magnetic resonance imaging (MRI) of the frontal and temporal, rTMS can suppress areas of cortical plasticity. This cortical reorganization can be demonstrated by magnetoencephalography (MEG)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic tinnitus
* Chronic subjective tinnitus for more than 6 months
* Pure tone average <50 dB HL in the ear where tinnitus is perceived
* Dominant tinnitus frequency measured between 4 and 8 kHz
* Subject is naive regarding rTMS
* Other concurrent treatments: A four-week washout from any other tinnitus
* treatment or management program is required prior to entering this study
* Stable enough to complete this study per the opinion of the Study Physician
* No restrictions, provided the dosages have been in place for at least 3 months
* A three month washout from any other tinnitus treatment or management program is required prior to entering this study.

Exclusion Criteria:

* Objective tinnitus or tinnitus with treatable cause
* Absolute thresholds > 60 dB on individual frequencies up to 8 kHz
* Presence of intracranial or intraocular ferromagnetic materiel or particles Cardiac pacemaker or other electronic implants (including cochlear implant)
* Serious heart disease or other unstable major medical condition

Personal history of central nervous system disorder, head injury, stroke or seizures

* Familial history of epilepsy;
* Concomitant medication with antidepressants and antipsychotics
* Pregnant women
* Severe depression
* Severe anxiety
* Others known contraindications to rTMS or brain MRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in MEG Asymmetry Index and amplitude of the auditory area | Baseline, After active treatment week

SECONDARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | Baseline, day 3, day 7, day 14, 1, 2 and 3 months after the first intervention
Visual Analog Scales (VAS) | Baseline, day 3, day 7, day 14, 1, 2 and 3 months after the first intervention
State-Trait Anxiety Inventory (STAI) | Baseline, before and after each intervention, 1, 2 and 3 months after the first intervention
Pittsburgh Sleep Quality Index (PSQI) | Baseline, before and after each intervention, 1, 2 and 3 months after the first intervention
Beck Depression Inventory (BDI) | Baseline, before and after each intervention, 1, 2 and 3 months after the first intervention

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Whan Suh, MD, ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Noh TS, Kyong JS, Park MK, Lee JH, Oh SH, Chung CK, Kim JS, Suh MW. Treatment Outcome of Auditory and Frontal Dual-Site rTMS in Tinnitus Patients and Changes in Magnetoencephalographic Functional Connectivity after rTMS: Double-Blind Randomized Controlled Trial. Audiol Neurootol. 2019;24(6):293-298. doi: 10.1159/000503134. Epub 2019 Dec 12. PMID 31830753